CLINICAL TRIAL: NCT00003384
Title: Expression of the MN Protein in Atypical Glandular Cells of Undetermined Significance (Agus or Agcus) As a Potential Diagnostic Biomarker of Cervical Dysplasia/Neoplasia
Brief Title: Protein Expression as a Potential Diagnostic Biomarker of Cervical Dysplasia and/or Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: GOG Foundation (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: GOG-171; NCI-2012-02269 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000066380; GOG-171 (Other: Gynecologic Oncology Group); GOG-0171 (Other: CTEP)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2015-05-29 (Estimated); Status verified 2015-05

CONDITIONS: Precancerous Condition; Stage 0 Cervical Cancer
MeSH Terms: conditions — Precancerous Conditions; Uterine Cervical Dysplasia | interventions — Vaginal Smears; Conization

ARMS (1):
- Diagnostic (Experimental): Patients undergo a Pap smear followed by a ThinPrep cervical cell specimen collection at the time of direct colposcopic examination. Patients then undergo a cone biopsy of the cervix using loop electrosurgical excision procedure with an endocervical curettage, an excisional cone biopsy of the cervix with or without endocervical curettage, or a hysterectomy. Patients who are perimenopausal or postmenopausal or have a negative cervical cone biopsy also undergo endometrial biopsy or curettage. The Pap smear specimen is analyzed to determine MN antigen expression and the ThinPrep specimen is analyzed for the presence of high-risk human papilloma virus and to determine MN antigen and other marker (e.g., P16) expression.
  Patients who do not undergo hysterectomy are followed every 6 months for 2 years. All other patients are followed at 4, 26, and 30 weeks.
  Interventions: Other: Cervical Papanicolaou Test; Procedure: Conization; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Other: Cervical Papanicolaou Test — Undergo Pap smear
  Other Names: Cervical Pap Test
Procedure: Conization — Undergo cone biopsy
  Other Names: cone biopsy; Cone Biopsy of Cervix; Conization of Cervix; Conization of Uterine Cervix
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This diagnostic trial is studying the presence of a specific protein as a potential biomarker of cervical dysplasia and/or cancer. The presence of specific proteins may allow a doctor to determine whether a patient has cervical dysplasia and/or cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Evaluate the utility of MN protein, a novel tumor-associated antigen, as a potential diagnostic biomarker for cervical glandular and/or squamous neoplasia in patients with a cytologic diagnosis of atypical glandular cells of undetermined significance (AGUS).

II. Measure the frequency and type of cervical pathology associated with the diagnosis of AGUS in these patients.

III. Determine whether the presence of a high-risk type of human papilloma virus (HPV) in a ThinPrep cervical cell specimen predicts the presence of cervical glandular and/or squamous cell neoplasia in these patients.

IV. Determine the relationship between MN antigen expression and the presence of high-risk HPV in these patients.

OUTLINE: This is a multicenter study.

Patients undergo a Pap smear followed by a ThinPrep cervical cell specimen collection at the time of direct colposcopic examination. Patients then undergo a cone biopsy of the cervix using loop electrosurgical excision procedure with an endocervical curettage, an excisional cone biopsy of the cervix with or without endocervical curettage, or a hysterectomy. Patients who are perimenopausal or postmenopausal or have a negative cervical cone biopsy also undergo endometrial biopsy or curettage. The Pap smear specimen is analyzed to determine MN antigen expression and the ThinPrep specimen is analyzed for the presence of high-risk human papilloma virus and to determine MN antigen and other marker (e.g., P16) expression.

Patients who do not undergo hysterectomy are followed every 6 months for 2 years. All other patients are followed at 4, 26, and 30 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Cytologically confirmed atypical glandular cells of undetermined significance (AGUS)
* Must be scheduled to undergo complete histologic examination of the cervix by cone biopsy using loop electrosurgical excision procedure with an endocervical curettage, excisional cone biopsy with or without endocervical curettage, or hysterectomy within 6 months of the initial cytologic diagnosis of AGUS
* No history of endometrial hyperplasia
* No history of cancer of the endometrium, vagina, or cervix
* HIV negative
* No pregnant patients who are at high risk for excessive bleeding or preterm labor if a cone biopsy is performed
* No prior cytotoxic chemotherapy for vaginal and/or cervical cancer
* No prior radiotherapy to the vagina or cervix
* No concurrent radiotherapy to the vagina or cervix
* No prior hysterectomy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 684 (Actual)
Dates: Start 1998-09; Primary Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Expression of the MN antigen in cytologic preparations that have been classified as AGUS | Baseline
Number of cervical specimens identified as having or not having glandular and/or squamous neoplasia | Baseline

SECONDARY OUTCOMES:
Ability of the MN antigen marker to be able to correctly predict patients who do not have glandular and/or squamous neoplasia | Up to 2 years
Feasibility, based on the number of years required to complete the study, as determined by both the actual disease prevalence rate as well as the actual patient accrual rate | At 1 year
Sensitivity for HIV testing | Baseline
Sensitivity of the expression of the MN antigen | Baseline
Specificity for HIV testing | Baseline
Specificity of the expression of the MN antigen | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Shu-Yuan Liao, Principal Investigator — Gynecologic Oncology Group
Locations (1):
- Gynecologic Oncology Group of Arizona, Phoenix, Arizona, United States